CLINICAL TRIAL: NCT00003327
Title: A Phase II Trial of Paclitaxel (TAXOL) Administered as a Weekly One Hour Infusion in Previously Treated Patients With Advanced Head and Neck Cancer
Brief Title: Paclitaxel in Treating Patients With Recurrent or Refractory Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066279; THERADEX-B97-5250; BMS-TAX/MEN.05; NCI-V98-1415
Record Dates: First submitted 1999-11-01; First posted 2004-03-22 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2001-11

CONDITIONS: Head and Neck Cancer
Keywords: stage IV nasopharyngeal cancer; recurrent nasopharyngeal cancer; stage IV lip and oral cavity cancer; recurrent lip and oral cavity cancer; stage IV hypopharyngeal cancer; recurrent hypopharyngeal cancer; stage IV laryngeal cancer; recurrent laryngeal cancer; stage IV paranasal sinus and nasal cavity cancer; recurrent paranasal sinus and nasal cavity cancer; stage IV oropharyngeal cancer; recurrent oropharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Nasopharyngeal Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients with recurrent or refractory head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate of paclitaxel as salvage therapy in patients with recurrent or refractory head and neck cancer. II. Evaluate the safety of paclitaxel in this patient population. III. Assess the overall survival and quality of life in these patients.

OUTLINE: This is an open label, multicenter, nonrandomized study. Patients receive intravenous paclitaxel over 1 hour weekly. Each course consists of four weeks. Patients receive treatment until disease progression or unacceptable toxic effects are observed. Patients are followed every 2 months for the first year, then every 4 months until completion of treatment, and then every 3 months until death. Patients complete a quality of life questionnaire prior to each of the first 6 courses, then every 2 courses thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or refractory head and neck cancer Measurable or evaluable disease At least one prior chemotherapy regimen for recurrent or metastatic disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL AST or ALT no greater than 2 times upper limit of normal (ULN) Renal: Creatinine no greater than 2 times ULN Calcium within normal limits Cardiovascular: No New York Heart Association class III-IV heart disease No myocardial infarction within 6 months No congestive heart failure No unstable angina No clinically significant pericardial effusions or arrhythmias Neurologic: No peripheral neuropathy greater than grade 1 Other: Not pregnant or nursing Fertile patients must use effective contraceptive method Negative pregnancy test No active infection or serious underlying medical condition No history of hypersensitivity to drugs containing Cremophor (teniposide, cyclosporine, or vitamin K) No prior invasive malignancies within the past 2 years, except: Curatively treated basal or squamous cell carcinoma of the skin Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior immunotherapy No concurrent immunotherapy Chemotherapy: See Disease Characteristics At least 5 weeks since prior nitrosoureas, melphalan, or mitomycin At least 3 weeks since other prior chemotherapy Prior taxane therapy allowed only if administered on a 3 week or greater schedule No concurrent chemotherapy Endocrine therapy: At least 3 weeks since prior hormonal therapy Concurrent megestrol (Megace) allowed No other concurrent hormonal therapy Radiotherapy: At least 3 weeks since prior radiotherapy No prior radiotherapy to greater than 30% of bone marrow No concurrent radiotherapy Surgery: At least 3 weeks since major surgery Other: At least 1 week since prior parenteral antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1997-09

CONTACTS AND LOCATIONS:
Overall Officials: Arlene A. Forastiere, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (20):
- United States (20):
  - California Cancer Center, Fresno, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Memorial Regional Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Savannah Hematology Oncology Associates, Savannah, Georgia
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Kansas City Internal Medicine, Kansas City, Missouri
  - Lourdes Regional Cancer Center, Binghamton, New York
  - Saint Vincent Catholic Medical Center of New York, New York, New York
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Medical Oncology Hematology Associates, Inc., Dayton, Ohio
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Cancer Care Institute of South Texas, San Antonio, Texas
  - Danville Hematology and Oncology, Inc., Danville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin